CLINICAL TRIAL: NCT03312972
Title: F-SHARP: A Phase I/II Trial of Focal Salvage High-dose-rate BRachytherapy for Locally Recurrent Prostate Cancer in Patients Treated With Prior Radiotherapy
Brief Title: Focal Salvage HDR Brachytherapy for Locally Recurrent Prostate Cancer in Patients Treated With Prior Radiotherapy
Acronym: F-Sharp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Abhishek A. Solanki, Assistant Professor of Radiation Oncology, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209557
Record Dates: First submitted 2017-09-22; First posted 2017-10-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Locally Recurrent Prostate Cancer
Keywords: Cancer; HDR Brachytherapy; Prostate Cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HDR Brachytherapy (Experimental): HDR Brachytherapy implant, Up to 30 Gray (Gy) to target lesion in one to two fractions.
  Interventions: Radiation: HDR Brachytherapy

INTERVENTIONS:
Radiation: HDR Brachytherapy — HDR Brachytherapy implant, deliver 1 to 2 fractions, Up to 30 Gray (Gy) to target lesion

SUMMARY:
This purpose of this study is to evaluate the safety and effectiveness of a technique called focal high-dose-rate (HDR) brachytherapy as treatment for prostate cancer that has come back in the prostate after prior radiotherapy. The study will examine the safety and efficacy of the treatment. The type of radiation that participants in this research will receive is targeted directly at the areas of the prostate where recurrent disease is evident, while avoiding treatment of the normal appearing prostate. This involves the placement of a radioactive material in the affected area of the prostate temporarily, where it remains for a short period of time, and then is subsequently removed using a minimally invasive technique called HDR Brachytherapy.

DETAILED DESCRIPTION:
The goal of any radiation treatment plan is to achieve maximal disease response with minimal toxicity. HDR brachytherapy offers a promising definitive treatment option in the setting of Locally Recurrent Prostate Cancer after prior definitive radiation, based on the limited data described above, with achievement of biochemical disease control in a large percentage of patients with relatively low toxicity. With focal HDR brachytherapy, the investigators can treat the isolated areas of disease, while avoiding normal prostate tissue, with the goal of further improving toxicity rates. The investigators hypothesize that using single fraction, focal HDR brachytherapy performed with one single implant for the treatment of LRPC is feasible and without excess toxicity, and can be safely delivered. This should allow for better patient convenience and cost and improved treatment dosimetry and planning, as it will decrease the risk of catheter displacement between fractions, which will hopefully correlate to less GU and non-GU acute toxicity. The primary objective is to determine the acute and late GU and GI toxicity of single fraction focal HDR salvage brachytherapy (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven locally recurrent adenocarcinoma of the prostate after the completion of definitive radiation therapy for initially diagnosed prostate cancer.

  * Biopsy must be performed within 182 days of trial registration
  * Biopsy should be a standard sextant biopsy AND either a targeted MR/ultrasound guided biopsy or saturation biopsy or both.
* Initial cancer diagnosis that fits these specific criteria:

  * Stages T1-T3a
  * Nx or N0
  * Mx or M0
* Eligible initial definitive radiotherapy modalities include:
* External beam radiotherapy, with photon or proton beam therapy

  * Conventional or moderately hypofractionated radiotherapy
  * Extremely hypofractionated external beam radiotherapy (Stereotactic body radiation therapy)
* Definitive Brachytherapy:

  * Low-dose rate
  * High-dose rate
* Locally recurrent disease confined to the prostate +/- seminal vesicles and immediately adjacent tissue, as evaluated by the following:

  * History/Physical examination
  * Radiographically node negative disease (N0), as defined by CT or MR of pelvis +/- abdomen within 6 months of registration.
  * No evidence of bone metastases (M0) on bone scan within 6 months of registration.
  * Fluciclovine-PET is encouraged, but not required
* Patients receiving ADT are eligible as long as they meet the other eligibility criteria. However, the duration of all ADT must be documented.
* Current ECOG Performance status Scale 0-2
* Current International Prostate Symptom Score (IPSS) < 20
* The patient must be medically suitable to receive general anesthesia.
* The patient must be able and willing to sign a study-specific written informed consent form before study entry.

Exclusion Criteria:

* Preregistration GI or GU toxicity (for any reason) grade ≥ 3 as defined in CTCAE version 4.03. That is, grade ≥ 3 GU or GI toxicity after first course of radiotherapy
* Patients receiving any other investigational agents.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, severely symptomatic congestive heart failure, cardiac arrhythmia, recent myocardial infarction in last 6 months, or psychiatric illness/social situations that could limit compliance with study requirements.
* Patients who have received chemotherapy or immunotherapy within one month prior to study enrollment, other than ADT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity rate | 24 months
  The primary outcome in this study is the number of acute or chronic grade 3-5 toxicities as described by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Solanki, MD, Principal Investigator — Loyola University
Locations (2):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Parekh A, Graham PL, Nguyen PL. Cancer control and complications of salvage local therapy after failure of radiotherapy for prostate cancer: a systematic review. Semin Radiat Oncol. 2013 Jul;23(3):222-34. doi: 10.1016/j.semradonc.2013.01.006. PMID 23763889
- [Background] Shipley WU, Thames HD, Sandler HM, Hanks GE, Zietman AL, Perez CA, Kuban DA, Hancock SL, Smith CD. Radiation therapy for clinically localized prostate cancer: a multi-institutional pooled analysis. JAMA. 1999 May 5;281(17):1598-604. doi: 10.1001/jama.281.17.1598. PMID 10235152
- [Background] Zelefsky MJ, Kuban DA, Levy LB, Potters L, Beyer DC, Blasko JC, Moran BJ, Ciezki JP, Zietman AL, Pisansky TM, Elshaikh M, Horwitz EM. Multi-institutional analysis of long-term outcome for stages T1-T2 prostate cancer treated with permanent seed implantation. Int J Radiat Oncol Biol Phys. 2007 Feb 1;67(2):327-33. doi: 10.1016/j.ijrobp.2006.08.056. Epub 2006 Nov 2. PMID 17084558
- [Background] Zumsteg ZS, Spratt DE, Romesser PB, Pei X, Zhang Z, Kollmeier M, McBride S, Yamada Y, Zelefsky MJ. Anatomical Patterns of Recurrence Following Biochemical Relapse in the Dose Escalation Era of External Beam Radiotherapy for Prostate Cancer. J Urol. 2015 Dec;194(6):1624-30. doi: 10.1016/j.juro.2015.06.100. Epub 2015 Jul 10. PMID 26165583
- [Background] Ahmadi H, Daneshmand S. Androgen deprivation therapy for prostate cancer: long-term safety and patient outcomes. Patient Relat Outcome Meas. 2014 Jul 5;5:63-70. doi: 10.2147/PROM.S52788. eCollection 2014. PMID 25045284
- [Background] Wirth MP, Hakenberg OW, Froehner M. Antiandrogens in the treatment of prostate cancer. Eur Urol. 2007 Feb;51(2):306-13; discussion 314. doi: 10.1016/j.eururo.2006.08.043. Epub 2006 Sep 11. PMID 17007995
- [Background] Grado GL, Collins JM, Kriegshauser JS, Balch CS, Grado MM, Swanson GP, Larson TR, Wilkes MM, Navickis RJ. Salvage brachytherapy for localized prostate cancer after radiotherapy failure. Urology. 1999 Jan;53(1):2-10. doi: 10.1016/s0090-4295(98)00492-0. PMID 9886580
- [Background] Beyer DC. Permanent brachytherapy as salvage treatment for recurrent prostate cancer. Urology. 1999 Nov;54(5):880-3. doi: 10.1016/s0090-4295(99)00241-1. PMID 10565751
- [Background] Skowronek J. Low-dose-rate or high-dose-rate brachytherapy in treatment of prostate cancer - between options. J Contemp Brachytherapy. 2013 Mar;5(1):33-41. doi: 10.5114/jcb.2013.34342. Epub 2013 Mar 29. PMID 23634153
- [Background] Grills IS, Martinez AA, Hollander M, Huang R, Goldman K, Chen PY, Gustafson GS. High dose rate brachytherapy as prostate cancer monotherapy reduces toxicity compared to low dose rate palladium seeds. J Urol. 2004 Mar;171(3):1098-104. doi: 10.1097/01.ju.0000113299.34404.22. PMID 14767279
- [Background] Yamada Y, Kollmeier MA, Pei X, Kan CC, Cohen GN, Donat SM, Cox BW, Zelefsky MJ. A Phase II study of salvage high-dose-rate brachytherapy for the treatment of locally recurrent prostate cancer after definitive external beam radiotherapy. Brachytherapy. 2014 Mar-Apr;13(2):111-6. doi: 10.1016/j.brachy.2013.11.005. Epub 2013 Dec 25. PMID 24373762
- [Background] Chen CP, Weinberg V, Shinohara K, Roach M 3rd, Nash M, Gottschalk A, Chang AJ, Hsu IC. Salvage HDR brachytherapy for recurrent prostate cancer after previous definitive radiation therapy: 5-year outcomes. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):324-9. doi: 10.1016/j.ijrobp.2013.01.027. Epub 2013 Mar 6. PMID 23474112
- [Background] Peters M, Maenhout M, van der Voort van Zyp JR, Moerland MA, Moman MR, Steuten LM, van Deursen MJ, van Vulpen M. Focal salvage iodine-125 brachytherapy for prostate cancer recurrences after primary radiotherapy: a retrospective study regarding toxicity, biochemical outcome and quality of life. Radiother Oncol. 2014 Jul;112(1):77-82. doi: 10.1016/j.radonc.2014.06.013. Epub 2014 Jul 3. PMID 24998704
- [Background] Sasaki H, Kido M, Miki K, Kuruma H, Takahashi H, Aoki M, Egawa S. Salvage partial brachytherapy for prostate cancer recurrence after primary brachytherapy. Int J Urol. 2014 Jun;21(6):572-7. doi: 10.1111/iju.12373. Epub 2013 Dec 23. PMID 24372730
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Derived] Solanki AA, Yoo RK, Adams W, Davicioni E, Mysz ML, Shea S, Gupta GN, Showalter T, Garant A, Hentz C, Farooq A, Baldea K, Small W, Harkenrider MM. F-SHARP: a Phase I/II trial of focal salvage high-dose-rate brachytherapy for Radiorecurrent prostate cancer. BJU Int. 2024 Feb;133(2):188-196. doi: 10.1111/bju.16150. Epub 2023 Sep 15. PMID 37562825